CLINICAL TRIAL: NCT00672204
Title: Efalizumab (Raptiva) Combined With Sirolimus in Type 1 Diabetic Islet Allograft Recipients
Brief Title: Raptiva and Sirolimus in Islet Transplantation for Type 1 Diabetes
Acronym: RAPTIVA
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Raptiva was withdrawn from the market
Sponsor: University of Minnesota (Other)
Collaborators: Juvenile Diabetes Research Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0612M98726
Record Dates: First submitted 2008-05-02; First posted 2008-05-06 (Estimated); Results first posted 2013-03-27 (Estimated); Last update posted 2017-10-25 (Actual); Status verified 2017-09

CONDITIONS: Type 1 Diabetes Mellitus; Hypoglycemia
Keywords: Islet transplant; Diabetes Mellitus; Hypoglycemia
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Hypoglycemia; Diabetes Mellitus | interventions — efalizumab; Sirolimus; Antilymphocyte Serum; thymoglobulin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): Allogeneic islets of Langerhans
  Interventions: Biological: Allogeneic islets of Langerhans transplant; Drug: Raptiva; Drug: Sirolimus; Drug: anti-thymocyte globulin

INTERVENTIONS:
Biological: Allogeneic islets of Langerhans transplant — Up to 3 intraportal infusions of cadaveric pancreatic islets of Langerhans. Each infusion to contain at least 5,000 islet equivalents/kg body weight.
  Other Names: Islets
Drug: Raptiva — Treatment Day -1 pretransplant to Treatment Day 90 after tx.: 1.0 mg/kg/wk SQ; Treatment Day 91 to Treatment Day 365: 0.5 mg/kg/wk SQ;
  Other Names: Efalizumab
Drug: Sirolimus — Initial dose 0.1 mg/kg PO on day -2, followed by 0.05 mg/kg daily, whole blood 24-hour trough adjusted to target 3-15 ng/ml as tolerated
  Other Names: Rapamune
Drug: anti-thymocyte globulin — 2.0 mg/kg on days -2, and -1 IV
  Other Names: ATG; Thymoglobulin

SUMMARY:
The primary objective of this protocol is to test the safety and efficacy of a treatment regimen consisting of maintenance therapy with efalizumab and sirolimus for 1 year followed by withdrawal of efalizumab and maintenance therapy with sirolimus, for the prevention of the destruction and rejection of islet transplants in type 1 diabetic recipients.

Genentech, the manufacturer of efalizumab voluntarily withdrew the drug from the U.S. market in April of 2009. Previously transplanted subjects have been transitioned to alternative immunosuppressives and no new subjects will be transplanted under this protocol.

DETAILED DESCRIPTION:
The purpose of this study is to improve the applicability of islet transplantation for treatment of type 1 diabetes utilizing a novel immunosuppressive regimen centered on the use of adhesion molecule blockade with an anti-LFA-1 antibody (efalizumab). The lymphocyte-function associated antigen-1 (LFA-1) adhesion molecule is expressed on multiple cellular populations including T cells, B cells, and NK cells and is important in facilitating cell migration and homing. In addition, interaction of LFA-1 with its ligand ICAM-1 on antigen presenting cells provides a powerful costimulatory signal for T cell activation.

Animal models using anti-LFA-1 antibodies have shown impressive prolongation of vascularized and cellular allograft survival. These potent immunosuppressive properties have also been documented in several clinical trials with efalizumab, a humanized IgG1 monoclonal antibody directed against LFA-1. The drug was found to be safe, well tolerated, and efficacious in treating moderate to severe psoriasis.

More recently, a multicenter trial employing efalizumab in conjunction with prednisone, sirolimus and cyclosporine maintenance immunosuppression in recipients of kidney allografts showed an acceptable safety profile when used at a dose of 0.5mg/kg/week and excellent rejection-free graft survival over the first 6 months after transplant.

This study represents the first clinical trial that applies adhesion molecule blockade with efalizumab to prevent the immune response against pancreatic islets in the setting of type 1 diabetes mellitus, with the long-term goal of immunosuppression withdrawal.

Genentech, the manufacturer of efalizumab voluntarily withdrew the drug from the U.S. market in April of 2009. Previously transplanted subjects have been transitioned to alternative immunosuppressives and no new subjects will be transplanted under this protocol.

ELIGIBILITY:
Inclusion Criteria:

1. Primary islet allotransplant
2. Type I diabetes mellitus for a minimum of 5 years
3. One of the following signs or symptoms despite intensive efforts made in close cooperation with their diabetic care team:

   * Metabolic lability/instability characterized by hypoglycemia or ketoacidosis (>2 hospital admissions in the previous year), erratic glucose profiles (MAGE>120 mg/dL), or disruption in lifestyle of danger to life, self or others
   * Reduced awareness of hypoglycemia or >1 episode in the last 1.5 years of severe hypoglycemia
   * Persistently poor glucose control (as defined by HgbA1c>10% at the end of six months of intensive management efforts with the diabetes care team)
   * Progressive secondary complications as defined by (i) a new diagnosis by an ophthalmologist of proliferative retinopathy or clinically significant macular edema or therapy with photocoagulation during the last year; or (ii) urinary albumin excretion rate >300 mg/day but proteinuria <3g/day; or (iii) symptomatic autonomic neuropathy (as defined by postural hypotension in the setting of euvolemia, gastroparesis or diarrhea attributed to diabetic neuropathy, or neuropathic bladder as diagnosed by an urologist)
4. Age 18 to 65 years of age.

Exclusion Criteria:

1. Current use of immunosuppressive agents
2. Lymphopenia (<1000/µL) or leukopenia (<3000 total leukocytes/µL)
3. Presence of panel-reactive anti-HLA antibody >20%
4. Positive lymphocytotoxic cross-match using donor lymphocytes and serum
5. Evidence of acute EBV infection (IgM>IgG) OR negative screen for EBV by IgG determination
6. Calculated or measured GFR < 60 ml/min/m2
7. Portal hypertension or history of significant liver disease
8. History of malignancy within 10 years (except for adequately treated basal or squamous cell CA of the skin)
9. Active peptic ulcer disease
10. Severe unremitting diarrhea or other GI disorders potentially interfering with the ability to absorb oral medications
11. Untreated proliferative retinopathy
12. Pregnancy or breastfeeding
13. Female subjects not post-menopausal or surgically sterile, or not using an acceptable method of contraception
14. Active infections
15. Serologic evidence of infection with HIV, or HbsAg or HCV Ab positive
16. Major ongoing psychiatric illness
17. Ongoing substance abuse, drug or alcohol; or recent history of noncompliance
18. Any condition that in the opinion of the Principle Investigator would not allow for safe participation in the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2007-11; Primary Completion 2010-12 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bernhard J. Hering, M.D., Principal Investigator — University of Minnesota
Locations (1):
- Universtiy of Minnesota, Minneapolis, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruited from 2008 - 2009 at the University of Minnesota.
Pre-assignment Details: Raptiva was removed from market.
Groups:
- Allogeneic Islets of Langerhans: Allogeneic islets of Langerhans
  anti-thymocyte globulin : 2.0 mg/kg on days -2, and -1 IV
  Raptiva : Treatment Day -1 pretransplant to Treatment Day 90 after tx.: 1.0 mg/kg/wk SQ; Treatment Day 91 to Treatment Day 365: 0.5 mg/kg/wk SQ;
  Allogeneic islets of Langerhans transplant : Up to 3 intraportal infusions of cadaveric pancreatic islets of Langerhans. Each infusion to contain at least 5,000 islet equivalents/kg body weight.
  Sirolimus : Initial dose 0.1 mg/kg PO on day -2, followed by 0.05 mg/kg daily, whole blood 24-hour trough adjusted to target 3-15 ng/ml as tolerated
Period: Overall Study
Arm/Group | Allogeneic Islets of Langerhans
Started | 23
Completed | 3
Not Completed | 20

BASELINE CHARACTERISTICS:
Arm/Group | Allogeneic Islets of Langerhans
Number analyzed (Participants) | 23
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 23
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.1 (9.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 8
Region of Enrollment [Number; unit: participants]
  United States | 23

OUTCOME MEASURES:

1. Primary Outcome: The Proportion of Insulin-independent Subjects With Full Islet Graft Function
Description: Islet transplant recipients will be considered insulin-independent with full islet graft function if they are able to titrate off insulin therapy for at least 1 week and all of the following criteria are met:
  * HbA1c < 7.0% or a ≥2.5% decrease from baseline;
  * fasting capillary glucose level should not exceed 140 mg/dL (7.8 mmol/L) more than three times in the past week (based on measuring capillary glucose levels a minimum of 7 times in a seven day period);
  * 2-hour post-prandial capillary glucose should not exceed 180 mg/dl (10.0 mmol/L) more than three times in the past week (based on measuring capillary glucose levels a minimum of 21 times in a seven day period);
  * fasting serum glucose level ≤126 mg/dL (7.0 mmol/L); if the fasting serum glucose level is >126 mg/dL (7.0 mmol/L), it must be confirmed in an additional one out of two measurements;
  * evidence of endogenous insulin production defined as fasting or stimulated C-peptide levels ≥0.5 ng/mL (0.16 nmol/L).
Time Frame: 1 year following the first islet transplant
Population: Raptiva was removed from market after 3 subjects were transplanted
Measure: Number; unit: participants
Arm/Group | Allogeneic Islets of Langerhans
Number analyzed (Participants) | 3
participants | 3

ADVERSE EVENTS:
Arm/Group | Allogeneic Islets of Langerhans
Serious Adverse Events (participants affected / at risk) | 0/3
Other Adverse Events (participants affected / at risk) | 0/3

LIMITATIONS AND CAVEATS:
Early termination due to Raptiva being withdrawn from market

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes